CLINICAL TRIAL: NCT01909258
Title: Comparison and Reproducibility of Pelvic Area Extension Measurements for Four Types of Lumbopelvic Balance Using Three Different Methods: Clinical Observation Versus Photography Versus the EOS Imaging System
Brief Title: Pelvic Area Extension Measurements for Four Types of Lumbopelvic Balance Using Three Different Methods
Acronym: CRESPEOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AOI/2012/PK; 2013-A00232-43 (Other: ANSM)
Record Dates: First submitted 2013-07-18; First posted 2013-07-26 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2016-05

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The study population. (Experimental): Healthy volunteers 20 to 40 years of age.
  Intervention: Goniometric measure of pelvic extension reserve. Intervention: Photographic measure of pelvic extension reserve. Intervention: EOS measure of pelvic extension reserve.
  Interventions: Other: Goniometric measure of pelvic extension reserve.; Other: Photographic measure of pelvic extension reserve.; Other: EOS measure of pelvic extension reserve.

INTERVENTIONS:
Other: Goniometric measure of pelvic extension reserve. — The pelvic extension reserve (°) is measured via goniometry.
  The goniometric measurements will be taken once by an investigator on all subjects and once by a different investigator on half of the subjects (with balanced distribution of morphotypes).
Other: Photographic measure of pelvic extension reserve. — The pelvic extension reserve (°) is measured using photography.
  Photographic measurements will be performed twice one investigator and 1 time by a different investigator (total of three measurements).
Other: EOS measure of pelvic extension reserve. — The pelvic extension reserve (°) is measured using the imaging system EOS.
  Five X-rays will be made for each volunteer on the EOS system. The first is a frontal shot in a bipedal position, reference snapshot for verifying the absence of spinal deformity or hip pathology. The second and third are profile shots, one on the left and one on the right, whole body, bipedal position; serving as a reference picture. The fourth is profile shot, whole body, with the left hip in hyperextension. For maximum left hip hyperextension, the right leg rests on a step of varying height, and the hip is maximally flexed. The fifth is a profile shot, full body, with the right hip in hyperextension. For a maximum right hip hyperextension, the left leg rests on a step of varying height, and the hip is maximally flexed.

SUMMARY:
The main objective of this study is to describe for the first time the expansion reserve of the pelvic area (measurements using the EOS system) for each of the four morphotypes (Roussouly classification) commonly found in a population of healthy volunteers.

DETAILED DESCRIPTION:
Secondary objectives:

A. The intra-judge reproducibility and the interrater reliability for the different tools used to measure hip extension will be evaluated. Intra-judge reproducibility (photography) and interrater reliability (goniometry and photography) for the different tools used for measuring hip extension will be evaluated.

B. The concordance between EOS measurements and measurements acquired via goniometry and photography will be evaluated.

C. Describe certain radiographic measurements via the EOS system for the four morphotypes

ELIGIBILITY:
Inclusion Criteria:

* The healthy volunteer must have given his/her informed and signed consent
* The healthy volunteer must be insured or beneficiary of a health insurance plan

Exclusion Criteria:

* The healthy volunteer is participating in another study
* The healthy volunteer is in an exclusion period determined by a previous study
* The healthy volunteer is under judicial protection, under tutorship or curatorship
* The healthy volunteer refuses to sign the consent
* It is impossible to correctly inform the healthy volunteer
* The healthy volunteer is pregnant, parturient, or breastfeeding
* The healthy volunteers had a history of chronic pain or surgery at the hip, the thoracolumbar spine or the sacroiliac area
* The healthy volunteer has a hip, knee or ankle abnormality

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04-25 (Actual); Study Completion 2016-04-25 (Actual)

PRIMARY OUTCOMES:
EOS measurement of intrinsic reserve extension = angular variation of the sacral slope (left and right sides) | baseline (day 0)
  = RIEeos
EOS measurement of extrinsic extension reserve | Baseline (day 0)
  = REEeos = angular variation of a specific angle (line joining the center of the sacral plate and the midpoint of the segment involving the center of the femoral head and the line joining this point to the top of the intercondylar knee notch) (left and right sides)
EOS measurement of global extension reserve | Baseline (day 0)
  = RIEeos + REEeos (left and right sides)

SECONDARY OUTCOMES:
Goniometric measurement of global extension reserve | baseline (day 0)
  (left and right sides)
Photographic measurement of global extension reserve | baseline (day 0)
  (left and right sides)
Roussouly classification: 1, 2, 3 or 4 | baseline (day 0)
Pelvic incidence (°) | Baseline (day 0)
  Pelvic Incidence is defined as the angle between two lines: the line perpendicular to the sacral endplate at the middle of the sacral endplate to the line between the middle of the sacral endplate to the middle of the femoral heads.
Standing sacral slope at rest | Baseline (day 0)
Standing sacral slope in extension | Baseline (day 0)
Standing pelvic tilt at rest | Baseline (day 0)
Standing pelvic tilt in extension | Baseline (day 0)
Standing anterior pelvic plane | Baseline (day 0)
The front acetabular inclination while standing | Baseline (day 0)
The sagittal acetabular inclination while standing | Baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Kouyoumdjian, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Kouyoumdjian P, Mansour J, Haignere V, Demattei C, Maury E, George D, Coulomb R. Hip-Spine Relationship between Sagittal Balance of the Lumbo-Pelvi-Femoral Complex and Hip Extension Capacity: An EOS Evaluation in a Healthy Caucasian Population. Global Spine J. 2024 Jan;14(1):265-271. doi: 10.1177/21925682221103831. Epub 2022 May 23. PMID 35604878